CLINICAL TRIAL: NCT03895190
Title: Effects of a Application (Flourish App) on Stress, Well-being and Emotional Regulation in Medical Students
Brief Title: Effects of a Application (Flourish App) in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HIAE_Florescer_Medicina
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-03

CONDITIONS: Emotional Stress
Keywords: well-being; stress; positive psychology; meditation; mobile application (app); medical students
MeSH Terms: conditions — Stress, Psychological; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control App (No Intervention): Initially this control group will have access to a Control App and after 8 weeks this goup will receive the intervention (Flourishing App Program).
- Experimental: Flourishing App Program (Experimental): This group will receive the intervention Flourishing App Program and after that it will not receive any other intervention.
  Interventions: Behavioral: Flourishing App Program

INTERVENTIONS:
Behavioral: Flourishing App Program — This intervention is based on relaxation, well-being promotion, meditation practices and positive psychology principles. The program is being evaluated in a classroom format into another project and was adapted for this project in the application format for mobile devices. It will last for 8 weeks, with trainings of 15 to 25 minutes, four times a week.
  Arms: Experimental: Flourishing App Program

SUMMARY:
This protocol proposes a well-being program, delivered through an application for mobile devices, based on meditation and positive psychology principles such as human development, the improvement of virtues, quality of life and well-being. The investigators hypothesize that this program offered in mobile application may promote well-being, reduce stress related problems and improving emotional regulation in the participants. Objectives: To evaluate the effectiveness of a well-being program delivered through an application for mobile devices in a sample of medical students. Methods: Three hundred students of the undergraduate medical course of Albert Einstein Israelite Faculty will be recruited. The participants will be randomized in two groups of 150 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI).

DETAILED DESCRIPTION:
INTRODUCTION: One population that presents an important vulnerability to stress is that of university students, facing several stressors, such as academic demands, time pressure and social adjustments. Medical students in particular may face additional challenges such as heavy workload, time commitment and the number of tests and assessments as well as the pressures of a clinical setting. Some highly successful programs in stress management are based on the principle of Mindfulness. On the other hand, Positive Psychology brings a new paradigm in terms of mental and emotional health, seeking to promote human development through the development of virtues, quality of life and well-being, instead of just treating disease. In the modern world not all people are willing to attend classroom training for several reasons. In this sense, a program offered in mobile application can be considered an interesting alternative for professionals that not only want to reduce stress-related symptoms, but also promote well-being.

MAIN OBJECTIVES: Evaluate the effects of a well-being program compared to a control program, both served on mobile applications, in reducing stress, increasing well-being and improving emotional regulation in a sample of medical students.

METHOD: For this purpose, 300 students of the undergraduate medical course of Albert Einstein Israelite Faculty. Participants will be randomized into groups of 150 each, half to the control group (CG) and the other half to the intervention group (IG). The IG will participate in the Flourish App Program, for 8 weeks, while the CG will have access to a control application. Then, after the evaluations, the CG will participate in the Flourish App Program, while the first group will not participate in any intervention. Before starting the program, after 4 and 8 weeks of the program, questions will be applied to assess the stress and well-being levels of participants in general and in relation to work. In addition, before and after each training period, questions will be applied to assess the stress and well-being levels of participants at the moment. Also, the Perceived Stress Scale, the 5-item World Health Organization Well-Being Index - WHO-5, the Mindful Attention Awareness Scale, the Self-Compassion Scale and the Difficulties in Emotion Regulation Scale will be applied too. Finally, at the end of the program, the Mobile Application Rating Scale - MARS will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Women and men from 17 years
* Students of the undergraduate medical course of Albert Einstein Israelite Faculty

Exclusion Criteria:

-

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Changes in subjective symptoms of well-being at work | baseline, 4 weeks, 8 weeks
  Sliding scale for stress level from 0 to 100
Changes in subjective symptoms of stress | baseline, 4 weeks, 8 weeks
  Sliding scale for well-being level from 0 to 100

SECONDARY OUTCOMES:
Changes in subjective symptoms of stress at the moment assessed using the sliding scale for stress | four times a week, before and after the period of each class (20 minutes)
  Sliding scale for stress level from 0 to 100
Changes in subjective symptoms of well-being at the moment assessed using the sliding scale for well-being | four times a week, before and after the period of each class (20 minutes)
  Sliding scale for well-being level from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Elisa H Kozasa, PhD, Principal Investigator — Instituto do Cérebro- Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil